CLINICAL TRIAL: NCT00915174
Title: Study to Evaluate the Effects of Neramexane on the Pharmacokinetics of a Combined Drospirenone/Ethinyl Estradiol Oral Contraceptive in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Manager Public Disclosure, Merz Pharmaceuticals GmbH
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: MRZ 92579/TI/1005
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2011-05

CONDITIONS: Healthy
Keywords: drug-drug interaction study
MeSH Terms: interventions — neramexane

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Neramexane — 25 mg q.d., 3 days 2 x 25 mg b.i.d., 11 days

SUMMARY:
Primary:

To assess the effects of repeated dose of Neramexane on the steady-state pharmacokinetics of Drospirenone [DRSP] and Ethinyl Estradiol [EE]

Secondary:

To assess safety and tolerability of concomitant repeated dose treatments of Neramexane and a fixed-combinational DRSP- and EE-containing oral contraceptive [OC] (Yasmin®)

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult female subject of child bearing potential (including subject with tubal ligation), white origin, who is able to read, to write and fully understand German language
* Aged 18 to 45 years (both inclusive)
* BMI of 18-28 kg/m2 and a body weight of 50-90 kg (both inclusive)
* The subject is required
* To have taken a DRSP/EE- containing OC for at least two dosing cycles
* To agree using reliable non hormonal birth control methods from Day -1 of study Period 1 until the Final Examination (e.g. non-hormonal IUD, double barrier method [e.g. condom with spermicide or diaphragm with spermicide], sexual abstinence). Women with tubal ligation or sterilized partner do not need an additional birth control method
* Willing and able to provide written informed consent after having been informed of the requirements and the restrictions of the study

Exclusion Criteria:

* History of clinically relevant allergy or known hypersensitivity to Neramexane/Memantine/ Amantadine and their derivatives
* Hypersensitivity to Quinine
* History of clinically relevant allergy or known hypersensitivity to any inactive ingredient in any of the used study medications (Neramexane, Yasmin®, Placebo) or tool substance
* History of clinically relevant allergy or known hypersensitivity to DRSP/EE
* Clinically relevant findings on the mammae or genital examination, PAP smear ≥ III
* Any contraindications against the oral contraceptive:
* present or past venous thromboses (deep vein thrombosis, pulmonary embolism);
* present or past arterial thromboses (e.g. myocardial infarction) or their prodromal stages (e.g. angina pectoris and transitory ischaemic attack);
* present or past cerebrovascular insult;
* presence of a serious risk factor or several risk factors for an arterial thrombosis: diabetes mellitus with vascular changes, severe hypertension, severe lipid metabolism disturbance;
* known or suspected genetic or acquired predisposition for venous or arterial thromboses like APC resistance,
* known or suspected genetic lack of antithrombin III, lack of protein C, lack of protein S, hyperhomocysteinaemia and antiphospholipid antibodies (anticardiolipin antibodies, lupus anticoagulants);
* present or past pancreatitis if this is accompanied by severe hypertriglyceridaemia;
* present or past severe hepatic disease as long as the liver function tests have not normalized;
* severe renal insufficiency or acute renal failure;
* present or past hepatic tumors (benign or malign);
* known or suspected sexual hormone dependent, malign tumors (e.g. of the genital organs or the mamma);
* diagnostic not clarified vaginal bleedings;
* anamnesis of migraine with focal neurologic symptoms;
* known hereditary angioedema
* Exposure to another investigational agent within the last two months before Day 1 of Period 1

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Area Under Curve within a dose interval (AUC, 0-tau) and Maximum Plasma Concentration at Steady State (Cmax) of Drospirenone (DRSP) and Ethinyl Estradiol (EE) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — Merz Pharmaceuticals
Locations (1):
- AAIharma Deutschland GmbH & Co. KG, Neu-Ulm, Bavaria, Germany